CLINICAL TRIAL: NCT02549092
Title: An Open-label, Randomized 26-Week Study Comparing Levodopa-Carbidopa INteStInal Gel (LCIG) THerapy to Optimized Medical Treatment (OMT) on Non-Motor Symptoms (NMS) in Subjects With Advanced Parkinson's Disease - INSIGHTS Study
Brief Title: A Study to Examine the Effect of Levodopa-Carbidopa Intestinal Gel (LCIG) Therapy Relative to That of Optimized Medical Treatment (OMT) on Non-motor Symptoms (NMS) Associated With Advanced Parkinson's Disease (PD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M12-927; 2014-004865-26 (EudraCT Number)
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Results first posted 2021-06-03 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Advanced Parkinson's Disease
Keywords: levodopa-carbidopa intestinal gel; levodopa; carbidopa; Advanced Parkinson's Disease; Non-Motor Symptom Scale NMSS; Parkinson's Disease Sleep Scale PDSS-2; efficacy
MeSH Terms: interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Optimized Medical Treatment (OMT) (Active Comparator): Participants randomized to continue OMT remain on their current optimized regimen. During the 26-week treatment phase, changes to anti-PD and NMS medications are to remain stable and can only be made if medically indicated.
  Eligible participants may elect to enter an extension/transition follow-up period to receive an individually optimized LCIG dose (after NJ and/or PEG-J placement), in order to transition to commercially available LCIG.
  Interventions: Drug: Optimized Medical Treatment; Drug: Levodopa-Carbidopa Intestinal Gel; Device: Nasojejunal (NJ) tube; Device: Percutaneous endoscopic gastrostomy with a jejunal (PEG-J) tube
- Levodopa-Carbidopa Intestinal Gel (LCIG) (Experimental): Participants randomized to LCIG at an individually optimized dose (after NJ and/or PEG-J placement), in accordance with the LCIG approved product label for countries participating in the study. During the 26-week treatment phase, changes to anti-PD and NMS medications are to remain stable and can only be made if medically indicated.
  The total daily dose of LCIG was composed of 3 components: (i) the morning dose, (ii) continuous maintenance infusion dose and (iii) extra doses. The continuous infusion is expected to run over a period of 16 consecutive hours each day.
  Eligible participants may elect to enter an extension/transition follow-up period to receive an individually optimized LCIG dose, in order to transition to commercially available LCIG.
  Interventions: Drug: Levodopa-Carbidopa Intestinal Gel; Device: Nasojejunal (NJ) tube; Device: Percutaneous endoscopic gastrostomy with a jejunal (PEG-J) tube

INTERVENTIONS:
Drug: Optimized Medical Treatment — Oral, sublingual or transdermal anti-PD medications and medications to treat NMS per Investigator discretion and/or in accordance with approved product label of the prescribed medications.
  Arms: Optimized Medical Treatment (OMT)
Drug: Levodopa-Carbidopa Intestinal Gel
  Other Names: ABT-SLV187; Duodopa; LCIG
Device: Nasojejunal (NJ) tube — optional prior to PEG-J placement
Device: Percutaneous endoscopic gastrostomy with a jejunal (PEG-J) tube

SUMMARY:
The primary objective of this study is to examine the effect of LCIG relative to that of OMT on NMS associated with PD.

DETAILED DESCRIPTION:
The study will consist of 3 sequential parts:

Part 1: Screening period. The screening period will consist of 3 visits, Visit 1 (V1), Visit 2 ([V2] [optional]) and the Randomization Visit (V3) in which the participant will be assessed to determine eligibility. The duration of the Screening Period can be between 30 to 67 days to accommodate the required procedures, training and collection of diaries, and to allow for stabilization of anti-PD medications and medications to treat NMS. All anti-PD medications and medications to treat NMS are required to be stable for a minimum of 30 days prior to randomization.

Part 2: Treatment period. Those participants randomized to OMT at the end of V3 will remain on their current optimized regimen. The day after randomization will be considered Day 1 of their treatment period and participants will have study visits at the end of Weeks 2, 6, 12, and 26. All participants randomized to the LCIG group should have all anti-PD medications, with the exception of levodopa formulations, tapered off within 14 days after randomization. Optional nasojujunal (NJ) and/or percutaneous endoscopic gastrostomy with a jejunal tube (PEG-J) placement will then occur. After that, the participant may begin initiation and titration of LCIG infusion to be adjusted to obtain the optimal clinical response. The day of initial NJ or PEG-J placement will be considered Day 1 for participants in the LCIG group. Study visits happen at the end of Weeks 2, 6, 12, and 26.

Part 3: Extension/Transition Period. Eligible participants who complete the 26 week study may continue into the Extension Period of the study. Participants in the LCIG arm will have study drug dispensation every 4 weeks and will have study visits every 6 months. Participants from the OMT arm will undergo the NJ (optional) and PEG-J procedures, titration, plus have visits at 2 weeks, 6 weeks, 3 months and 6 months post NJ or PEG-J. Participants will then continue to receive study drug every 4 weeks and will have study visits every 6 months until Duodopa is commercially available. Transition to a Post-Trial Access protocol will be possible if Duodopa does not become commercially available in a location.

ELIGIBILITY:
Inclusion Criteria:

1. Participant(s) must have a diagnosis of idiopathic Parkinson's disease according to the United Kingdom Parkinson's Disease Society (UKPDS) Brain Bank Criteria.
2. Participant(s) demonstrates persistent motor fluctuations in spite of individually optimized treatment.
3. The participant's Parkinson's disease is levodopa-responsive.
4. Participant(s) has had optimized treatment with available anti-PD medication and their motor symptoms are judged inadequately controlled on this optimized treatment. Optimized treatment is defined as the maximum therapeutic effect obtained with pharmacological antiparkinsonian therapies when no further improvement is expected regardless of any additional manipulations of levodopa and/or other antiparkinsonian medication. This will be based on the Investigator's clinical judgment.
5. Male or female participant(s) must be at least 30 years of age.
6. Minimum Parkinson's Disease Sleep Scale 2 (PDSS-2) total score of 18 at Baseline assessment.

Exclusion Criteria:

1. Participant's PD diagnosis is unclear or there is a suspicion that the subject has a parkinsonian syndrome such as secondary parkinsonism (e.g. caused by drugs, toxins, infectious agents, vascular disease, trauma, brain neoplasm), parkinson-plus syndrome (e.g. Multiple System Atrophy, Progressive supranuclear Palsy, Diffuse Lewy Body disease) or other neurodegenerative disease that might mimic the symptoms of PD.
2. Participant(s) has undergone neurosurgery for the treatment of Parkinson's disease.
3. Known hypersensitivity to levodopa, carbidopa or radiopaque material.
4. Participant(s) has contraindications to levodopa (e.g. narrow angle glaucoma, malignant melanoma).
5. Participant(s) experiencing clinically significant sleep attacks or clinically significant impulsive behavior (e.g. pathological gambling, hypersexuality) at any point during the three months prior to the Screening evaluation as judged by the Principal Investigator.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (38):
- United States (8):
  - Parkinson's and Movement /ID# 161596, Fountain Valley, California
  - Boca Raton Regional Hospital /ID# 200056, Boca Raton, Florida
  - University of Florida Neurolog /ID# 168699, Jacksonville, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida /ID# 168085, Port Charlotte, Florida
  - Rush University Medical Center /ID# 168088, Chicago, Illinois
  - St. Luke's Health System /ID# 168706, Kansas City, Missouri
  - Central Texas Neurology Consul /ID# 168087, Round Rock, Texas
  - Inland Northwest Research /ID# 200113, Spokane, Washington
- Australia (4):
  - Westmead Hospital /ID# 136575, Westmead, New South Wales
  - Royal Adelaide Hospital /ID# 136577, Adelaide, South Australia
  - Royal Melbourne Hospital /ID# 136780, Parkville, Victoria
  - Goulburn Valley Hospital /ID# 164202, Shepparton, Victoria
- Canada (3):
  - University of Alberta /ID# 136586, Edmonton, Alberta
  - The Ottawa Hospital /ID# 139341, Ottawa, Ontario
  - Toronto Western Hospital /ID# 136585, Toronto, Ontario
- Central Hospital Bremerhaven /ID# 136573, Bremerhaven, Germany
- Greece (2):
  - 251 Airforce General Hospital /ID# 160594, Athens, Attica
  - Mediterraneo Hospital /ID# 208042, Glyfada
- Italy (7):
  - A.O. Univ. Ospedali Riuniti /ID# 135964, Ancona, The Marches
  - Ospedale Bellaria.Azienda USL IRCCS.Istituto delle Scienze Neurologiche di Bolog /ID# 136789, Bologna
  - A.O.U. Ospedali Riuniti di Fog /ID# 136792, Foggia
  - A.O.U. Policlinico G. Martino /ID# 136790, Messina
  - Ospedale S.Maria della Miseri /ID# 160609, Perugia
  - Azienda Sanitaria Locale di /ID# 160608, Ponderano,biella
  - Azienda Policlinico Umberto I /ID# 201223, Roma
- South Korea (3):
  - Severance Hospital /ID# 163019, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 162990, Seoul
  - Asan Medical Center /ID# 163018, Seoul
- Spain (9):
  - Hospital Universitario de Bellvitge /ID# 136579, L'Hospitalet de Llobregat, Barcelona
  - CHU Insular-Materno Infantil /ID# 136783, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Clinic de Barcelona /ID# 137689, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 136581, Barcelona
  - Hospital Puerta del Mar /ID# 157977, Cadiz
  - Hospital Universitario Virgen de las Nieves /ID# 136583, Granada
  - Hospital Universitario Ramon y Cajal /ID# 136784, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 145624, Seville
  - Hospital Universitario y Politecnico La Fe /ID# 136722, Valencia
- Karolinska Univ Sjukhuset /ID# 135961, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 32 sites in 9 countries.
Pre-assignment Details: After a 30- to 67-day Screening Period for required procedures, training, and medication stabilization, eligible participants were randomized to Optimized Medical Treatment (OMT) or Levodopa-Carbidopa Intestinal Gel (LCIG) for a 26-week Treatment Period. Before Treatment Period Day 1, LCIG participants had a percutaneous endoscopic gastrostomy with a jejunal extension (PEG-J; with an initial, optional, temporary nasojejunal [NJ] tube placement to titrate the dose of LCIG prior to the PEG-J).
Groups:
- Optimized Medical Treatment: Participants randomized to continue OMT remained on their current optimized regimen during the 26-week treatment phase. Changes to anti-PD and NMS medications are to remain stable and can only be made if medically indicated.
  Participants in the United States or South Korea may have elected to enter an Extension/Transition follow-up period to receive an individually optimized LCIG dose (after NJ and/or PEG-J placement), in order to transition to commercially available LCIG.
- LCIG: Participants randomized to LCIG at an individually optimized dose, in accordance with the LCIG approved product label for countries participating in the study during the 26-week treatment phase. Changes to anti-PD and NMS medications were to remain stable and were only made if medically indicated.
  The total daily dose of LCIG was composed of 3 components: (i) the morning dose, (ii) continuous maintenance infusion dose and (iii) extra doses. The continuous infusion was expected to run over a period of 16 consecutive hours each day.
  Participants in the United States or South Korea may have elected to enter an Extension/Transition follow-up period to receive an individually optimized LCIG dose, in order to transition to commercially available LCIG.
Period: Treatment Period
Arm/Group | Optimized Medical Treatment | LCIG
Started (Randomized) | 44 | 45
Completed (Completed 26-week Treatment Period) | 41 | 38
Not Completed | 3 | 7
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lack of Efficacy | 0 | 2
Period: Extension/Transition Period
Arm/Group | Optimized Medical Treatment | LCIG
Started | 10 | 14
Transitioned to Commercial LCIG | 5 | 7
Completed | 5 | 10
Not Completed | 5 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other, Not Specified | 4 | 2

BASELINE CHARACTERISTICS:
Population: Safety dataset: all participants randomized to OMT, and all participants randomized to LCIG who had study device (NJ and/or PEG-J) placement.
Groups:
- Total: Total of all reporting groups
Arm/Group | Optimized Medical Treatment | LCIG | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (6.21) | 66.9 (7.34) | 67.8 (6.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 14 | 34
  Male | 24 | 29 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 35 | 36 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 35 | 34 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Non-Motor Symptoms Scale (NMSS) Total Score [Mean (Standard Deviation); unit: score on a scale] — The NMSS consists of 30 questions in 9 domains (cardiovascular/falls, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastrointestinal (GI) tract, urinary, sexual function, miscellaneous). Score of each question is calculated by multiplying severity*frequency. Severity and frequency are rated using a scale ranging from 0 (none) to 3 (severe) for severity and from 1 (rarely) to 4 (very frequent) for frequency. Total score is the sum of 9 domains, and ranges from 0 to 360, with a lower value indicating a more desirable outcome. Population: Intent-to-Treat Data Set: all participants randomized to the OMT arm, and all participants randomized to LCIG arm who received at least one dose of study drug. Participants with a baseline measurement are reported in this table.
  score on a scale
    number analyzed (Participants) | 43 | 42 | 85
    (all) | 112.4 (51.37) | 99.7 (46.49) | 106.2 (49.14)
Modified Parkinson's Disease Sleep Scale (PDSS-2) Total Score [Mean (Standard Deviation); unit: score on a scale] — The PDSS-2 addresses PD-specific sleep disturbances such as restless leg syndrome (RLS), morning akinesia, pain, and sleep apnea. The frequency is assessed for the 15 sleep problems based on a 5-point Likert-type scale (ranging from 0 [never] to 4 [very often]). Scores are calculated for each of the 3 domains (motor symptoms at night, PD symptoms at night, and disturbed sleep) as well as a total score. The PDSS-2 domain scores range from 0 to 20 and the total score is a sum of the 3 domains and ranges from 0 to 60. Population: Intent-to-Treat Data Set: all participants randomized to the OMT arm, and all participants randomized to LCIG arm who received at least one dose of study drug. Participants with a baseline measurement are reported in this table.
  score on a scale
    number analyzed (Participants) | 43 | 42 | 85
    (all) | 30.3 (8.55) | 29.9 (7.36) | 30.1 (7.94)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in the NMSS Total Score
Description: The NMSS consists of 30 questions in 9 domains (cardiovascular/falls, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, GI tract, urinary, sexual function, miscellaneous). Score of each question is calculated by multiplying severity*frequency. Severity and frequency are rated using a scale ranging from 0 (none) to 3 (severe) for severity and from 1 (rarely) to 4 (very frequent) for frequency. Total score is the sum of 9 domains, and ranges from 0 to 360, with a lower value indicating a more desirable outcome. Repeated-measure analysis.
Time Frame: Baseline, Week 26
Population: Intent-to-Treat Data Set: all participants who were randomized to the OMT arm, and all participants who were randomized to LCIG arm and received at least one dose of study drug. Participants with baseline and a post-baseline measurement are reported in this table.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Optimized Medical Treatment: Participants randomized to continue OMT remained on their current optimized regimen during the 26-week treatment phase. Changes to anti-PD and NMS medications are to remain stable and can only be made if medically indicated.
- LCIG: Participants randomized to LCIG at an individually optimized dose, in accordance with the LCIG approved product label for countries participating in the study during the 26-week treatment phase. Changes to anti-PD and NMS medications were to remain stable and were only made if medically indicated.
  The total daily dose of LCIG was composed of 3 components: (i) the morning dose, (ii) continuous maintenance infusion dose and (iii) extra doses. The continuous infusion was expected to run over a period of 16 consecutive hours each day.
Arm/Group | Optimized Medical Treatment | LCIG
Number analyzed (Participants) | 43 | 42
score on a scale | -23.83 (8.30) | -32.04 (8.53)
Statistical Analysis 1: Comparison: Optimized Medical Treatment vs LCIG; Test type: Superiority; p = 0.410, mixed model repeated measures — P value is from the mixed model repeated measures (MMRM) with the model: change from Baseline=treatment, country, visit, Baseline, treatment-by-visit, and Baseline-by-visit. Unstructured variance-covariance structure was used in the MMRM analysis; Adjusted for multiplicity using the Hochberg procedure to control the family-wise error rate at a pre-specified significance level (alpha = 0.05); Least Squares (LS) Mean of Difference = -8.21, 95% CI 2-sided [-27.98 to 11.55], Standard Error of Mean 9.91 — Difference of LCIG - OMT

2. Primary Outcome: Change From Baseline to Week 26 in the Modified PDSS-2 Total Score
Description: The PDSS-2 addresses PD-specific sleep disturbances such as restless leg syndrome (RLS), morning akinesia, pain, and sleep apnea. The frequency is assessed for the 15 sleep problems based on a 5-point Likert-type scale (ranging from 0 [never] to 4 [very often]). Scores are calculated for each of the 3 domains (motor symptoms at night, PD symptoms at night, and disturbed sleep) as well as a total score. The PDSS-2 domain scores range from 0 to 20 and the total score is a sum of the 3 domains and ranges from 0 to 60. Repeated measure analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Optimized Medical Treatment | LCIG
Number analyzed (Participants) | 43 | 42
score on a scale | -8.98 (2.00) | -7.41 (2.01)
Statistical Analysis 1: Comparison: Optimized Medical Treatment vs LCIG; Test type: Superiority; p = 0.509, mixed model repeated measures — The P value is from the MMRM with the model: change from Baseline = treatment, country, visit, Baseline, treatment-by-visit, and Baseline-by-visit. The unstructured variance-covariance structure was used in the MMRM analysis; [statistical method as in outcome 1, analysis 1]; LS Mean of Difference = 1.57, 95% CI 2-sided [-3.16 to 6.30], Standard Error of Mean 2.37 — Difference of LCIG - OMT

3. Secondary Outcome: Change From Baseline to Week 26 in Parkinson's Disease Questionnaire (PDQ-8) Summary Index Score
Description: The PDQ-8 is a disease-specific instrument designed to measure aspects of health relevant to PD. Eight questions including the mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort are assessed on a 5-point scale: 0 = Never, 1 = Occasionally, 2 = Sometimes, 3 = Often, 4 = Always (or cannot do at all, if applicable). Summary index score is the sum of each question divided by 32 and multiplied by 100. Scores range from 0 to 100 with lower values desirable.
Time Frame: Baseline, Week 26
Population: Intent-to-Treat Data Set: all participants who were randomized to the OMT arm, and all participants who were randomized to LCIG arm and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Optimized Medical Treatment | LCIG
Number analyzed (Participants) | 44 | 43
score on a scale | -1.75 (2.96) | -5.56 (2.97)
Statistical Analysis 1: Comparison: Optimized Medical Treatment vs LCIG; Statistical significance for the 3 key secondary efficacy endpoints (PDQ-8 index score, CGI-C score, and UPDRS Part II) could only be evaluated using the Hochberg procedure for multiplicity control if both primary endpoints had been statistically significant after multiplicity adjustment; Test type: Superiority; p = 0.291, Repeated measures model — The repeated measures model: change = treatment, country, visit, baseline, treatment * visit, baseline * visit. The unstructured variance-covariance structure is used; LS mean difference = -3.81, 95% CI 2-sided [-10.96 to 3.34], Standard Error of Mean 3.59 — Difference of LCIG - OMT

4. Secondary Outcome: Clinical Global Impression of Change (CGI-C) Final Score
Description: CGI-C score is a clinician's impression of a subject's change in status on a 7-point scale (1 = very much improved, 2 = much improved, 3 = minimally Improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse). Scores range from 1 to 7, with lower score desirable.
Time Frame: End of Treatment Period (up to Week 26)
Population: Intent-to-Treat Data Set: all participants who were randomized to the OMT arm, and all participants who were randomized to LCIG arm and received at least one dose of study drug. Participants with an assessment are reported in this table.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Optimized Medical Treatment | LCIG
Number analyzed (Participants) | 43 | 40
score on a scale | 4.9 (0.25) | 2.5 (0.24)
Statistical Analysis 1: Comparison: Optimized Medical Treatment vs LCIG; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA — Analysis of covariance (ANCOVA) model: FINAL = treatment, country; LS Mean of Difference = -2.3, 95% CI 2-sided [-2.84 to -1.82], Standard Error of Mean 0.26 — Difference of LCIG - OMT

5. Secondary Outcome: Change From Baseline at Week 26 in Unified Parkinson's Disease Rating Scale (UPDRS) Part II Score
Description: UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's disease of 42 total questions. Part I (Questions 1 - 4), Part II (Questions 5 - 17), Part III (Questions 18 - 31), and Part IV (Questions 32 - 42). Questions 35 - 38 and 40 - 42 are 2-point (0 and 1), all other questions are 5-point (0 - 4). Part II scores range from 0 to 52 with lower value desirable.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Optimized Medical Treatment | LCIG
Number analyzed (Participants) | 44 | 43
score on a scale | 0.53 (0.89) | -2.26 (0.87)
Statistical Analysis 1: Comparison: Optimized Medical Treatment vs LCIG; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.006, Repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -2.79, 95% CI 2-sided [-4.77 to -0.81], Standard Error of Mean 0.99 — Difference of LCIG - OMT

6. Secondary Outcome: Change From Baseline to Week 26 in the NMSS Domain Scores
Description: The NMSS consists of 30 questions in 9 domains. Score of each question is calculated by multiplying severity*frequency. Severity and frequency are rated using a scale ranging from 0 (none) to 3 (severe) for severity and from 1 (rarely) to 4 (very frequent) for frequency. Cardiovascular/falls scores range from 0 - 24 with lower value desirable. Sleep/fatigue scores range from 0 - 48 with lower value desirable. Mood/cognition scores range from 0 - 72 with lower value desirable. Perceptual problems/hallucinations scores range from 0 - 36 with lower value desirable. Attention/memory scores range from 0 - 36 with lower value desirable. Gastrointestinal tract scores range from 0 - 36 with lower value desirable. Urinary scores range from 0 - 36 with lower value desirable. Sexual function scores range from 0 - 24 with lower value desirable. Miscellaneous scores range from 0 - 48 with lower value desirable. Repeated-measure analysis.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Optimized Medical Treatment | LCIG
Number analyzed (Participants) | 43 | 42
score on a scale
  Cardiovascular including falls | -1.84 (0.82) | -1.76 (0.86)
  Sleep/fatigue | -7.11 (2.02) | -6.06 (2.06)
  Mood/cognition | -5.99 (3.06) | -7.84 (3.11)
  Perceptual problems/hallucinations | -1.53 (0.70) | -1.14 (0.72)
  Attention/memory | -1.20 (1.60) | -2.15 (1.66)
  Gastrointestinal tract | -0.85 (1.09) | -3.43 (1.14)
  Urinary | -3.65 (1.90) | -4.83 (1.96)
  Sexual function | 0.88 (0.86) | 0.10 (0.90)
  Miscellaneous | -3.87 (1.53) | -5.16 (1.60)
Statistical Analysis 1: Comparison: Optimized Medical Treatment vs LCIG; Cardiovascular including falls; Test type: Superiority; p = 0.933, Repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS mean difference = 0.08, 95% CI 2-sided [-1.89 to 2.06], Standard Error of Mean 0.99 — Difference of LCIG - OMT
Statistical Analysis 2: Comparison: Optimized Medical Treatment vs LCIG; Sleep/fatigue; Test type: Superiority; p = 0.655, Repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS mean difference = 1.05, 95% CI 2-sided [-3.63 to 5.74], Standard Error of Mean 2.35 — Difference of LCIG - OMT
Statistical Analysis 3: Comparison: Optimized Medical Treatment vs LCIG; Mood/cognition; Test type: Superiority; p = 0.616, Repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -1.85, 95% CI 2-sided [-9.18 to 5.48], Standard Error of Mean 3.67 — Difference of LCIG - OMT
Statistical Analysis 4: Comparison: Optimized Medical Treatment vs LCIG; Perceptual problems/hallucinations; Test type: Superiority; p = 0.645, Repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS mean difference = 0.39, 95% CI 2-sided [-1.30 to 2.08], Standard Error of Mean 0.84 — Difference of LCIG - OMT
Statistical Analysis 5: Comparison: Optimized Medical Treatment vs LCIG; Attention/memory; Test type: Superiority; p = 0.645, Repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -0.94, 95% CI 2-sided [-5.03 to 3.14], Standard Error of Mean 2.04 — Difference of LCIG - OMT
Statistical Analysis 6: Comparison: Optimized Medical Treatment vs LCIG; Gastrointestinal tract; Test type: Superiority; p = 0.058, Repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -2.58, 95% CI 2-sided [-5.25 to 0.09], Standard Error of Mean 1.34 — Difference of LCIG - OMT
Statistical Analysis 7: Comparison: Optimized Medical Treatment vs LCIG; Urinary; Test type: Superiority; p = 0.588, Repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -1.18, 95% CI 2-sided [-5.52 to 3.15], Standard Error of Mean 2.17 — Difference of LCIG - OMT
Statistical Analysis 8: Comparison: Optimized Medical Treatment vs LCIG; Sexual function; Test type: Superiority; p = 0.464, Repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -0.78, 95% CI 2-sided [-2.88 to 1.33], Standard Error of Mean 1.05 — Difference of LCIG - OMT
Statistical Analysis 9: Comparison: Optimized Medical Treatment vs LCIG; Miscellaneous; Test type: Superiority; p = 0.468, Repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS mean difference = -1.29, 95% CI 2-sided [-4.80 to 2.23], Standard Error of Mean 1.76 — Difference of LCIG - OMT

7. Secondary Outcome: Change From Baseline to Week 26 in the Modified PDSS-2 Domain Scores
Description: as for outcome 2
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Optimized Medical Treatment | LCIG
Number analyzed (Participants) | 43 | 42
score on a scale
  Motor symptoms at night | -2.21 (1.04) | -2.79 (1.05)
  PD symptoms at night | -1.77 (0.66) | -1.53 (0.69)
  Disturbed sleep | -4.88 (0.74) | -2.89 (0.75)
Statistical Analysis 1: Comparison: Optimized Medical Treatment vs LCIG; Motor symptoms at night; Test type: Superiority; p = 0.643, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.58, 95% CI 2-sided [-3.09 to 1.92], Standard Error of Mean 1.26 — Difference of LCIG - OMT
Statistical Analysis 2: Comparison: Optimized Medical Treatment vs LCIG; PD symptoms at night; Test type: Superiority; p = 0.769, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = 0.24, 95% CI 2-sided [-1.39 to 1.87], Standard Error of Mean 0.82 — Difference of LCIG - OMT
Statistical Analysis 3: Comparison: Optimized Medical Treatment vs LCIG; Disturbed sleep; Test type: Superiority; p = 0.020, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = 1.99, 95% CI 2-sided [0.32 to 3.66], Standard Error of Mean 0.84 — Difference of LCIG - OMT

8. Secondary Outcome: Change From Baseline at Week 26 in UPDRS Parts I, III, and IV Score
Description: UPDRS is an investigator-used rating tool to follow the longitudinal course of Parkinson's disease of 42 total questions. Part I (Questions 1 - 4), Part II (Questions 5 - 17), Part III (Questions 18 - 31), and Part IV (Questions 32 - 42). Questions 35 - 38 and 40 - 42 are 2-point (0 and 1), all other questions are 5-point (0 - 4). Part I is the sum of Questions 1 - 4; scores range from 0 to 16 with lower value desirable. Part III is the sum of Questions 18 - 31 (Questions 20 - 26 apply to multiple body parts, resulting in 27 answers total); scores range from 0 to 108 with lower value desirable. Part IV is the sum of Questions 32 - 42; scores range from 0 to 23 with lower value desirable.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Optimized Medical Treatment | LCIG
Number analyzed (Participants) | 44 | 43
score on a scale
  Part I | 0.20 (0.39) | 0.39 (0.39)
  Part III: number analyzed (Participants) | 43 | 43
  Part III | 1.32 (1.84) | -0.89 (1.80)
  Part IV | -0.61 (0.53) | -2.31 (0.52)
Statistical Analysis 1: Comparison: Optimized Medical Treatment vs LCIG; Part I score; Test type: Superiority; p = 0.672, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = 0.19, 95% CI 2-sided [-0.72 to 1.10], Standard Error of Mean 0.46 — Difference of LCIG - OMT
Statistical Analysis 2: Comparison: Optimized Medical Treatment vs LCIG; Part III score; Test type: Superiority; p = 0.302, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -2.22, 95% CI 2-sided [-6.47 to 2.04], Standard Error of Mean 2.13 — Difference of LCIG - OMT
Statistical Analysis 3: Comparison: Optimized Medical Treatment vs LCIG; Part IV score; Test type: Superiority; p = 0.007, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -1.70, 95% CI 2-sided [-2.91 to -0.48], Standard Error of Mean 0.61 — Difference of LCIG - OMT

9. Secondary Outcome: Change From Baseline at Week 26 in Parkinson's Anxiety Scale (PAS) Total Score
Description: PAS is a 12-item scale developed specifically to measure severity in anxiety in Parkinson's disease for the following items: Feeling anxious or nervous; Feeling tense or stressed; Being unable to relax; Excessive worrying about everyday matters; Fear of something bad, or even the worst, happening; Panic or intense fear; Shortness of breath; Heart palpitations or heart beating fast; Fear of losing control; Social situations; Public settings; Specific objects or situations. Severity for each item is rated as: 0, Never; 1 Rarely; 2, Sometimes; 3, Often; 4, Nearly always. Total score is the sum of the12 item scores, with a range of 0 to 48; a lower value is desirable.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Optimized Medical Treatment | LCIG
Number analyzed (Participants) | 44 | 41
score on a scale | -0.75 (1.28) | -2.29 (1.27)
Statistical Analysis 1: Comparison: Optimized Medical Treatment vs LCIG; Test type: Superiority; p = 0.307, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -1.54, 95% CI 2-sided [-4.52 to 1.44], Standard Error of Mean 1.50 — Difference of LCIG - OMT

10. Secondary Outcome: Change From Baseline at Week 26 in Geriatric Depression Scale (GDS-15) Score
Description: The GDS-15 is a short, self-report reliable and valid screening instrument for depression in the elderly of 15 yes/no questions: 1) Satisfied with life 2) Dropped many activities and interests 3) Life is empty 4) Often get bored 5) In good spirits most of the time 6) Afraid that something bad is going to happen 7) Feel happy most of the time 8) Often feel helpless 9) Prefer to stay at home, rather than going out and doing things 10) Feel that have more problems with memory than most 11) Think it is wonderful to be alive now 12) Feel worthless 13) Feel full of energy 14) Situation is hopeless 15) Most subjects are better off. Answers of 'yes' to questions 2, 3, 4, 6, 8, 9, 10, 12, 14, 15 are scored 1 point. Answers of 'no' to questions 1, 5, 7, 11, 13 are scored
  1 point. The 15 items are summed and scores range from 0 - 15 with lower value desirable.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Optimized Medical Treatment | LCIG
Number analyzed (Participants) | 44 | 43
score on a scale | 0.25 (0.40) | 0.17 (0.39)
Statistical Analysis 1: Comparison: Optimized Medical Treatment vs LCIG; Test type: Superiority; p = 0.868, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.08, 95% CI 2-sided [-0.99 to 0.84], Standard Error of Mean 0.46 — Difference of LCIG - OMT

11. Secondary Outcome: Change From Baseline at Week 26 in King's PD Pain Scale (KPPS) Score
Description: The KPPS score is a clinical PD-specific pain scale of 14 items addressing the following 7 domains: musculoskeletal pain, chronic pain, fluctuation-related pain, nocturnal pain, orofacial pain, neuropathic pain, radicular pain. Each domain item is scored by severity (0, none to 3, very severe) multiplied by frequency (0, never to 4, all the time) resulting in a subscore of 0 - 12 (with lower value desirable), the sum of the 14 items gives the total score with a range from 0 to 168 with lower value desirable.
Time Frame: Baseline, Week 26
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Optimized Medical Treatment | LCIG
Number analyzed (Participants) | 44 | 43
score on a scale
  Total score | -11.32 (2.83) | -12.46 (2.77)
  Musculoskeletal Pain Score | -1.72 (0.63) | -1.79 (0.62)
  Chronic pain score | -0.84 (0.54) | -0.77 (0.55)
  Fluctuation related pain score | -3.77 (1.30) | -3.14 (1.28)
  Nocturnal pain score | -2.41 (1.04) | -2.78 (1.01)
  Orofacial pain score | -0.74 (0.41) | -0.87 (0.41)
  Discoloration and edema score | -0.47 (0.65) | -2.27 (0.65)
  Radicular pain score | -1.43 (0.39) | -1.47 (0.39)
Statistical Analysis 1: Comparison: Optimized Medical Treatment vs LCIG; Total score; Test type: Superiority; p = 0.728, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -1.14, 95% CI 2-sided [-7.68 to 5.39], Standard Error of Mean 3.28 — Difference of LCIG - OMT
Statistical Analysis 2: Comparison: Optimized Medical Treatment vs LCIG; Musculoskeletal pain score; Test type: Superiority; p = 0.916, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.08, 95% CI 2-sided [-1.50 to 1.35], Standard Error of Mean 0.71 — Difference of LCIG - OMT
Statistical Analysis 3: Comparison: Optimized Medical Treatment vs LCIG; Chronic pain score; Test type: Superiority; p = 0.919, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = 0.07, 95% CI 2-sided [-1.28 to 1.42], Standard Error of Mean 0.68 — Difference of LCIG - OMT
Statistical Analysis 4: Comparison: Optimized Medical Treatment vs LCIG; Fluctuation related pain score; Test type: Superiority; p = 0.680, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = 0.63, 95% CI 2-sided [-2.42 to 3.68], Standard Error of Mean 1.53 — Difference of LCIG - OMT
Statistical Analysis 5: Comparison: Optimized Medical Treatment vs LCIG; Nocturnal pain score; Test type: Superiority; p = 0.767, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.37, 95% CI 2-sided [-2.83 to 2.09], Standard Error of Mean 1.24 — Difference of LCIG - OMT
Statistical Analysis 6: Comparison: Optimized Medical Treatment vs LCIG; Orofacial pain score; Test type: Superiority; p = 0.804, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.13, 95% CI 2-sided [-1.15 to 0.90], Standard Error of Mean 0.51 — Difference of LCIG - OMT
Statistical Analysis 7: Comparison: Optimized Medical Treatment vs LCIG; Discoloration and edema score; Test type: Superiority; p = 0.025, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -1.81, 95% CI 2-sided [-3.38 to -0.23], Standard Error of Mean 0.79 — Difference of LCIG - OMT
Statistical Analysis 8: Comparison: Optimized Medical Treatment vs LCIG; Radicular pain score; Test type: Superiority; p = 0.930, repeated measures model — [p-value comment as in outcome 3, analysis 1]; LS Mean of Difference = -0.04, 95% CI 2-sided [-0.99 to 0.90], Standard Error of Mean 0.47 — Difference of LCIG - OMT

12. Secondary Outcome: Patient Global Impression of Change (PGIC) Final Score
Description: The PGIC is a 7-point response scale. The participant was asked by the Investigator or qualified designee to rate their change in status using the following 7-point scale: 1 = Very much improved, 2 = Much improved, 3 = Minimally improved, 4 = No change, 5 = Minimally worse, 6 = Much worse, 7 = Very much worse. PGIC score ranges from 1 to 7 with lower score desirable.
Time Frame: End of Treatment Period (up to Week 26)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Optimized Medical Treatment | LCIG
Number analyzed (Participants) | 43 | 40
score on a scale | 4.9 (0.25) | 2.5 (0.24)
Statistical Analysis 1: Comparison: Optimized Medical Treatment vs LCIG; Test type: Superiority; p < 0.001, ANCOVA — ANCOVA model: FINAL = treatment, country; LS Mean of Difference = -2.4, 95% CI 2-sided [-2.89 to -1.87], Standard Error of Mean 0.26 — Difference of LCIG - OMT

ADVERSE EVENTS:
Time Frame: All adverse events are reported from the time of randomization until 30 days following last OMT dose, last study visit, discontinuation of study drug administration, removal of the PEG-J tube or Last LCIG Commercial Transition Visit have elapsed. Median duration of follow-up was 191 days for OMT and 565 days for LCIG in the Treatment Period, and was 1366 days for OMT -> LCIG and 1003.5 days for LCIG -> LCIG in the Extension/Transition period.
Groups:
- Optimized Medical Treatment (OMT): Participants randomized to continue OMT remained on their current optimized regimen during the 26-week treatment phase. Changes to anti-PD and NMS medications are to remain stable and can only be made if medically indicated.
- Extension/Transition OMT->LCIG: Participants randomized to continue OMT in the United States or South Korea who elected to enter an Extension/Transition follow-up period to receive an individually optimized LCIG dose (after NJ and/or PEG-J placement), in order to transition to commercially available LCIG.
- Extension/Transition LCIG->LCIG: Participants randomized to LCIG in the United States or South Korea who elected to enter an Extension/Transition follow-up period to receive an individually optimized LCIG dose, in order to transition to commercially available LCIG.
Arm/Group | Optimized Medical Treatment (OMT) | LCIG | Extension/Transition OMT->LCIG | Extension/Transition LCIG->LCIG
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/45 | 1/10 | 0/14
Serious Adverse Events (participants affected / at risk) | 4/44 | 9/43 | 2/10 | 1/14
Other Adverse Events (participants affected / at risk) | 13/44 | 33/43 | 6/10 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimized Medical Treatment (OMT) (N=44) | LCIG (N=43) | Extension/Transition OMT->LCIG (N=10) | Extension/Transition LCIG->LCIG (N=14)
AORTIC VALVE STENOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMOPERITONEUM (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERITONITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STOMA SITE INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Optimized Medical Treatment (OMT) (N=44) | LCIG (N=43) | Extension/Transition OMT->LCIG (N=10) | Extension/Transition LCIG->LCIG (N=14)
CATARACT NUCLEAR (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NORMAL TENSION GLAUCOMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 5 (6) | 1 (1) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRIC MUCOSAL LESION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
ASYMPTOMATIC COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STOMA SITE CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STOMA SITE INFECTION (Infections and infestations) | 0 (0) | 5 (5) | 1 (2) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 7 (8) | 4 (6) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
STOMA SITE DERMATITIS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STOMA SITE DISCHARGE (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
STOMA SITE HYPERGRANULATION (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (2) | 0 (0)
STOMA SITE PAIN (Injury, poisoning and procedural complications) | 0 (0) | 6 (7) | 3 (6) | 1 (1)
VITAMIN B6 DECREASED (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
DYSKINESIA (Nervous system disorders) | 1 (1) | 4 (4) | 2 (2) | 0 (0)
FREEZING PHENOMENON (Nervous system disorders) | 3 (4) | 1 (2) | 0 (0) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 3 (3) | 2 (3) | 0 (0) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEVICE DISLOCATION (Product Issues) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
DEVICE MALFUNCTION (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
IMPULSE-CONTROL DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
IMPULSIVE BEHAVIOUR (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 4 (4) | 1 (2) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SLEEP ATTACKS (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
SOCIAL PROBLEM (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT02549092/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT02549092/SAP_001.pdf